CLINICAL TRIAL: NCT06108141
Title: Implementation of a Novel Virtual Reality Intervention to Support Clinicians' Firearm Safety Counseling Behaviors
Brief Title: Virtual Reality Intervention to Support Clinicians' Firearm Safety Counseling Behaviors
Acronym: REACH_CCTST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, F. Joseph Real, Associate Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-0469
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Virtual Reality; Simulation Based Medical Education; Firearm Injury
Keywords: Virtual Reality; Simulation Based Medical Education; Firearm Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resident Education And Counseling on Household (REACH) Firearm Safety (Experimental): Resident participants will complete a modified online self-guided American Academy of Pediatrics (AAP) Safer curriculum. Next, residents will complete REACH individually with a trained facilitator.
  Interventions: Behavioral: Resident Education And Counseling on Household Firearm Safety
- Modified AAP Safer (Active Comparator): Resident participants will complete a modified online self-guided American Academy of Pediatrics (AAP) Safer curriculum.
  Interventions: Behavioral: Modified American Academy of Pediatrics Safer

INTERVENTIONS:
Behavioral: Resident Education And Counseling on Household Firearm Safety — An intervention that includes a self-directed online curriculum and virtual reality simulations, designed to teach firearm screening and counseling among clinicians.
  Other Names: REACH Firearm Safety
  Arms: Resident Education And Counseling on Household (REACH) Firearm Safety
Behavioral: Modified American Academy of Pediatrics Safer — An intervention that includes a self-directed online curriculum.
  Other Names: Modified AAP Safer
  Arms: Modified AAP Safer

SUMMARY:
The goal of this clinical trial is to assess the efficacy of REACH Firearm Safety in a sample of pediatric residents. The main question it aims to answer are:

Do residents who have completed REACH Firearm Safety have increased documentation in the electronic medical records for screening and counseling for safe firearm storage?

Participants will be asked to engage in a virtual reality curriculum (REACH Firearm Safety). Researchers will compare the REACH Firearm safety group to a group of participants who complete an abbreviated online training.

DETAILED DESCRIPTION:
The American Academy of Pediatrics urges pediatricians to counsel parents on the dangers of childhood access to firearms and restrict access through safe storage practices. However, evidence suggests that most pediatricians do not provide firearm-related counseling in real-world clinical practice. This is notable as firearm-related injury is now the leading cause of death in children aged 1-19 years in the United States. Virtual reality (VR) is a type of simulation-based medical education that allows users to interact with virtual environments and characters in a seemingly realistic way. Investigators developed Resident Education And Counseling on Household (REACH) Firearm Safety, a VR curriculum to allow pediatricians to practice screening and counseling on firearm safety. The objective of this proposal is to assess the efficacy of REACH Firearm Safety, along with key implementation metrics, to justify and inform scale and distribution of the training approach. To achieve the objective, Investigators will: (1) Conduct a multi-site two-arm randomized controlled pilot study assessing the efficacy of REACH Firearm Safety and (2) Measure acceptability, appropriateness, fidelity, feasibility, and cost of implementation of REACH Firearm Safety. The proposed research is significant and innovative because it is the first rigorous effort to evaluate the efficacy of VR as a training platform to teach communication skills related to firearm safety counseling.

ELIGIBILITY:
Inclusion Criteria:

* Resident with continuity clinic at either Kentucky Clinic South, University of Kentucky (UK) Internal Medicine and Pediatrics group, CCHMC Hopple Street Neighborhood Health Center, or University of Cincinnati (UC) Hoxworth Medicine-Pediatrics Clinic

Exclusion Criteria:

* Resident unable to read or speak English
* Resident with continuity clinic outside of inclusion criteria clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in the Percentage of Participants with documentation within the medical record of access to firearms. | 6 months
  Documentation of discussion during clinical encounter of access to firearms.
Percent Change From Baseline in the Percentage of Participants with documentation within the medical record of counseling on firearm injury prevention. | 6 months
  Documentation of discussion during clinical encounter of firearm injury prevention.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No